CLINICAL TRIAL: NCT02539238
Title: The Effect of a New Training Program on CPR Quality of Pediatric Healthcare Providers: A Randomized Control Trial With Economic Evaluation
Brief Title: Improving CPR Quality With Longitudinal Practice and Realtime Feedback - RCT With CEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Yiqun Lin, MD, MHSc, PhD candidate, Simulation Fellow, Alberta Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: REB14-1352
Record Dates: First submitted 2015-08-23; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Medical Education; cardiopulmonary resuscitation; feedback; cost-effectiveness analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): Annual BLS training
  Interventions: Other: Longitudinal practice and real-time feedback
- intervention (Experimental): Brief CPR training dispersed over a year period of time with real-time feedback during working hour
  Interventions: Other: Longitudinal practice and real-time feedback

INTERVENTIONS:
Other: Longitudinal practice and real-time feedback — Brief CPR practice distributed during working hours with real-time feedback

SUMMARY:
Objectives: The primary objective of this project is to assess whether the implementation of a new cardiopulmonary resuscitation (CPR) training program (longitudinal training with real-time feedback) can improve CPR quality of healthcare providers compared with traditional training method. The secondary objective is to identify whether the implementation of the new training program will result in cost-effectiveness.

Design: Randomized trial to compare new training program with tradition training method and cost-effectiveness alongside this trial

Participants and setting: Paediatric healthcare providers in Emergency Department at Alberta Children's Hospital. Subjects will be enrolled in either intervention (new training program) or control (traditional training program) by random.

Statistical analysis: Investigators will conduct chi-square test and independent t-test to compare the proportion of excellent CPR and 3 metrics of CPR quality of intervention group with control group at the end of 12-month interval. A multi-level logistic regression and linear regression models will be used to assess the effect of training method and time on proportion of excellent CPR and 3 metrics of CPR quality. Investigators will also conduct a full-economic evaluation in a health care system prospective. cost-effectiveness will be expressed as cost per increased CPR excellence according to incremental cost-effectiveness ratio (ICER). A one-way sensitivity analysis and a probabilistic sensitivity analysis will be conducted to deal with uncertainty in effects and costs.

Conclusion: The new CPR training program will serve as an example of competency-based psychomotor skill training program and help healthcare providers to improve quality of CPR, and potentially improve the survival of children with cardiac arrest. The results of the studies might provide evidence to inform and update in resuscitation education guideline to change the way of CPR training and improve the cost-effectiveness of CPR training program.

DETAILED DESCRIPTION:
The study utilizes a randomized, paralleled study design.Paediatric healthcare providers (nurses and physicians) will be enrolled into one of two arms: (1) longitudinal just-in-time training with real-time feedback (intervention); or (2) Annual BLS recertification course (control).

Participants and Setting: The study will be conducted in the Emergency Department (ED) at Alberta Children's Hospital (ACH), a paediatric tertiary care and referral center in Calgary, Alberta, Canada. Annual BLS recertification courses are organized for healthcare providers in the emergency department every month and all healthcare providers in ED are scheduled to take the course once each year. The investigators will approach potential participants and seek consent from them during the course.

Intervention: longitudinal just-in-time training with real-time feedback The new CPR training curriculum (longitudinal just-in-time training with real-time feedback) provides on-demand CPR training opportunities in a longitudinal fashion with a continuous flow of practice, assessment, and feedback. Each CPR training station has a cart with an adult/paediatric sized CPR torso manikin and an infant manikin. The training unit also includes a real-time visual feedback device to provide quality of CPR feedback (depth, rate, and recoil of compressions) during compressions (referred to as real time feedback). At the end of each CPR practice event, the unit will provide summative feedback for the learner on the quality of CPR (depth, rate, recoil and overall quality). Health care providers in our study will have easy access to the training units, which will be located in the emergency department (ED) simulation lab. The instructional process consists of 2 parts, practice sessions and assessment sessions.

Each day, healthcare providers assigned to the ED resuscitation room for their clinical shift will practice CPR for 2 minutes with real-time feedback (if they are enrolled in the intervention arm of the study). Participants will do 2 minutes of continuous chest compressions while assuming that the patient is intubated. Training will take place in the ED simulation lab (located in the ED), a short 20-second walk from the resuscitation room. Providers will be encouraged to use the training unit each time they are on a resuscitation shift, but they will also have access to the training unit if they are not on a resuscitation shift. All health care providers in the intervention arm are recommended to attend practice sessions at least once a week, with no maximum for the number of times they are permitted to practice. After each practice session, participants will be presented with a quantitative summary of CPR performance (depth, rate, residual leaning force). Each training session will last approximately 3 minutes: 30 seconds for reviewing guidelines (short video), 2 minutes of CPR practice, 30 seconds for the participant to review their summative data. In order to encourage participants to practice, the investigators ask permission from ED administration to offer 5 minute protected time after hand-over of each shift and a research assistant will record times of practice for each participants enrolled in intervention group.

Assessment sessions will be built into the instruction framework of the intervention. The assessment session will be given at baseline and every 3 months over the course of one year. Assessment sessions will be run in the same setting as practice sessions. Subjects in will be expected to complete assessment sessions at baseline, 3, 6, 9, and 12 months intervals. Each participant will have protected time (after weekly rounds) for assessment sessions. During the assessment sessions:

1. Real time CPR feedback will not be available to all participants. Data will be collected for analysis only.
2. Participants will be presented with the quantitative summary of CPR performance only, if enrolled in the intervention arm.

Study Design: At the beginning of the study, both groups will undergo annual Basic Life Support (BLS) recertification training to ensure good CPR skill acquisition at baseline. All participants who provide consent will be recruited and randomized into one of the 2 study arms. The nurse educator, who is not a member of study group, will generate allocation sequence with an online random number generator. Given the attributes of the study, we will not be able to blind the participants or investigators.

Participants in both arms will be assessed after BLS recertification course as baseline assessment. The baseline assessment includes a CPR competency test and demographic information . Participants randomized to the intervention arm will participate in longitudinal just-in-time training with real-time feedback program as described above. Participants randomized to the control arm will undergo the current standard program of annual BLS recertification but will not participate in the interventional training program during the course of the year. Quantitative measures of CPR quality (compression depth, rate, recoil and overall performance) will be captured for all assessment sessions (in both intervention and control arm) at 3,6,9 and 12 months. For the control group, a second recertification course will be conducted at 1 year, after which CPR performance will be assessed in the same way. In order to ensure compliance, course instructors will send a reminder email to all participants for assessment, and they will be given some protected time (i.e. academic half day) for participating assessment sessions. The assessment sessions will take place in the Emergency Department simulation lab at Alberta Children's Hospital. Control group participants will be advised not to use the training unit for intervention group for CPR practice during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric Healthcare providers in the Emergency Department at Alberta Children's Hospital (nurses and physicians)

Exclusion Criteria:

* Not Basic Life Support (BLS), Advanced Cardiovascular Life Support (ACLS), or Pediatric Advanced Life Support (PALS) certified within the past two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Achieving "excellent CPR" at the end of the study (number and percentage) | month 12
  dichotomous variable based on chest compression depth, rate and recoil

SECONDARY OUTCOMES:
Change of percentage of adequate compression depth from baseline (numeric, percent) | month 3,6,9,12
  Percentage of chest compression with depth greater than 50 mm
Change of percentage of adequate compression rate from baseline (numeric, percent) | month 3,6,9,12
  Percentage of chest compression with rate between 100-120 per minute
Change of percentage of adequate compression recoil from baseline (numeric, percent) | month 3,6,9,12
  Percentage of chest compression with fully recoil between compressions

OTHER OUTCOMES:
Cost (Canadian Dollar) | month 12
  Cost of running both control and experimental educational program

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital/KidSIM simulation center, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Lin Y, Savage T, Gravel G, Davidson J, Tofil N, Duff J, Cheng A. Who is the real team leader? Comparing leadership performance of the team leader and CPR Coach during simulated cardiac arrest. Resusc Plus. 2023 May 24;14:100400. doi: 10.1016/j.resplu.2023.100400. eCollection 2023 Jun. PMID 37265710
- [Derived] Cheng A, Kessler D, Lin Y, Tofil NM, Hunt EA, Davidson J, Chatfield J, Duff JP; International Network for Simulation-based Pediatric Innovation, Research and Education (INSPIRE) CPR Investigators. Influence of Cardiopulmonary Resuscitation Coaching and Provider Role on Perception of Cardiopulmonary Resuscitation Quality During Simulated Pediatric Cardiac Arrest. Pediatr Crit Care Med. 2019 Apr;20(4):e191-e198. doi: 10.1097/PCC.0000000000001871. PMID 30951004
- [Derived] Lin Y, Cheng A, Grant VJ, Currie GR, Hecker KG. Improving CPR quality with distributed practice and real-time feedback in pediatric healthcare providers - A randomized controlled trial. Resuscitation. 2018 Sep;130:6-12. doi: 10.1016/j.resuscitation.2018.06.025. Epub 2018 Jun 23. PMID 29944894
- See also: KidSIM Simulation Research Program — http://www.kidsim.ca